CLINICAL TRIAL: NCT00930982
Title: Randomized, Placebo-controlled, Double-blind, Multi-center Study to Evaluate the Safety and Efficacy of Ciprofloxacin Inhale Compared to Placebo in Patients With Non-cystic Fibrosis Bronchiectasis
Brief Title: Evaluation of Cipro Inhale in Patients With Non-cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12965; 2009-009869-34 (EudraCT Number)
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-11

CONDITIONS: Bronchiectasis
Keywords: Ciprofloxacin; Airway infection; Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciprofloxacin Inhale (BAYQ3939) (Experimental): 32.5 mg ciprofloxacin hydrated corresponding to 50 mg Ciprofloxacin PulmoSphere Inhalation Powder twice daily
  Interventions: Drug: Ciprofloxacin (Cipro, BAYQ3939)
- Placebo (Placebo Comparator): Inhalation of matching placebo twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin (Cipro, BAYQ3939) — Inhalation of 32,5mg Ciprofloxacin inhaled twice a day
  Arms: Ciprofloxacin Inhale (BAYQ3939)
Drug: Placebo — Inhalation of matching placebo twice a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if bacterial load in the airways can be reduced after inhalation of ciprofloxacin for 28 days.

DETAILED DESCRIPTION:
Safety issues are addressed in the AE section. There is no standardised and unanimously accepted definition of exacerbation in COPD; 4 definitions are widely used: (1) using a combination of 3 cardinal symptoms: increased dyspnea, sputum volume, and sputum purulence; (2) looking at the presence of the following patterns of symptoms during >=2 consecutive days: either 2 or more of 3 major symptoms (increase in dyspnoea, sputum volume and sputum purulence); or any 1 major symptom together with any 1 minor symptom (increase in nasal discharge, wheeze, sore throat, cough or fever); (3) a sustained worsening of the patient's condition, from the stable state and beyond normal day-to-day variations, that is acute in onset and necessitates a change in regular medication in a patient with underlying COPD; (4) a complex of respiratory events (i.e. cough, wheezing, dyspnoea or sputum production) lasting >=3 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a proven and documented diagnosis of non-cystic fibrosis idiopathic or post pneumonic bronchiectasis
* Stable pulmonary status and stable regimen of standard treatment at least for the past 30 days

Exclusion Criteria:

* Forced Expiratory Volume 1 < 35% or > 80%
* Allergic bronchopulmonary aspergillosis
* Immunodeficiency disease requiring immunoglobulin replacement
* Inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (42):
- United States (11):
  - Little Rock, Arkansas
  - La Jolla, California
  - Denver, Colorado
  - Farmington, Connecticut
  - Washington D.C., District of Columbia
  - Naples, Florida
  - Michigan City, Indiana
  - Mineola, New York
  - Houston, Texas
  - Tyler, Texas
  - Payson, Utah
- Australia (7):
  - Concord, New South Wales
  - South Brisbane, Queensland
  - Woollongabba, Queensland
  - Adelaide, South Australia
  - Heidelberg, Victoria
  - Prahran, Victoria
  - Nedlands, Western Australia
- Germany (12):
  - Löwenstein, Baden-Wurttemberg
  - Rüdersdorf, Brandenburg
  - Frankfurt am Main, Hesse
  - Gelnhausen, Hesse
  - Hanover, Lower Saxony
  - Witten, North Rhine-Westphalia
  - Koblenz, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Geesthacht, Schleswig-Holstein
  - Großhansdorf, Schleswig-Holstein
  - Berlin, State of Berlin
  - Bad Berka, Thuringia
- Spain (4):
  - Santiago de Compostela, A Coruña
  - Badajoz, Badajoz
  - Barcelona, Barcelona
  - Palma de Mallorca, Illes Baleares
- Uppsala, Sweden
- United Kingdom (7):
  - Bristol, Avon
  - Cambridge, Cambridgeshire
  - Liverpool, Merseyside
  - Belfast, North Ireland
  - Newcastle upon Tyne, Tyne and Wear
  - Edinburgh
  - Norwich

REFERENCES:
- [Result] Wilson R, Welte T, Polverino E, De Soyza A, Greville H, O'Donnell A, Alder J, Reimnitz P, Hampel B. Ciprofloxacin dry powder for inhalation in non-cystic fibrosis bronchiectasis: a phase II randomised study. Eur Respir J. 2013 May;41(5):1107-15. doi: 10.1183/09031936.00071312. Epub 2012 Sep 27. PMID 23018904
- See also: Click here and search for Bayer products information provided by EMA — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pulmonary stable participants with a proven and documented diagnosis of non-cystic fibrosis bronchiectasis (idiopathic or postpneumonic), and on a stable regimen of standard treatment, were recruited at specialized study sites.
Pre-assignment Details: Out of 277 participants screened, 153 failed screening (mostly due to not meeting in-/exclusion criteria or inability to produce adequate sputum samples), and 124 participants were randomized (60 to Ciprofloxacin Inhale and 64 to placebo).
Period: Overall Study
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Started | 60 | 64
Completed | 39 | 35
Not Completed | 21 | 29
Not completed — Adverse Event | 19 | 23
Not completed — Protocol Violation | 1 | 5
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo | Total
Number analyzed (Participants) | 60 | 64 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (11.8) | 61.4 (11.9) | 63.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 43 | 82
  Male | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Bacterial Load in the Sputum at End of Treatment (Day 29).
Description: Total bacterial load was determined in sputum collected before the inhalation of study drug. Sputum samples were either provided by the participant during the respective study visit, or participants had to bring a sputum sample that had been produced within the 4 hours prior to the visit. Induced sputum samples could be collected if the participant was unable to produce a spontaneously expectorated sputum sample of > 2 mL. Imputation method: last observation carried forward (LOCF). CFU: colony forming units, log10: decadic logarithm
Time Frame: Baseline and 29 days
Population: Modified intent-to-treat (ITT) analyses were performed on all participants who had been randomized and received study drug. This population was identical to the ITT population of all randomized participants.
Measure: Mean (Standard Deviation); unit: log10 of CFU per gram sputum
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
log10 of CFU per gram sputum | -2.94 (3.40) | -0.32 (2.29)
Statistical Analysis 1: Comparison: Ciprofloxacin Inhale (BAYQ3939) vs Placebo; Ho: CFU(EOT|Cipro) - CFU(baseline|Cipro) > CFU(EOT|Placebo) - CFU(baseline|Placebo) CFU = colony forming units EOT=End of treatment (Day 29) Sample size was based a difference of 1.2 log10 CFU/g between placebo and Ciprofloxacin and a standard deviation of 2 log10 CFU/g; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value should be < 0.023 (one-sided) for a significant result as an interim analysis was performed. Results based on the no-interaction model which was defined as primary analysis; Baseline cfu was covariate, treatment and pooled centers factors. As the p-value for interaction was 0.214, the no-interaction model is appropriate; Difference in Least square means = -2.368, Standard Error of Mean 2.674 — Least square mean Ciprofloxacin minus placebo

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: Pulmonary function testing (spirometry) was conducted in accordance with American Thoracic Society standards. FEV1 was defined as the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration, expressed in liters at body temperature and ambient pressure saturated with water vapor (BTPS). Imputation method: last observation carried forward (LOCF).
Time Frame: Baseline and up to end of study (planned at Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of predicted FEV1
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
Percent of predicted FEV1
  Day 8 | -0.67 (4.50) | -0.14 (5.10)
  Day 29 | -0.53 (7.88) | -0.22 (9.57)
  Day 42 | 1.19 (5.88) | -0.26 (9.88)
  Day 56 | 0.81 (5.50) | -0.24 (9.61)
  Day 84 | 0.70 (5.69) | -0.50 (7.62)

3. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: Pulmonary function testing (spirometry) was conducted in accordance with American Thoracic Society standards. FVC was defined as the maximal volume of air exhaled with maximally forced effort from a maximal inspiration, i.e. vital capacity performed with a maximally forced expiratory effort expressed in liters at BTPS. Imputation method: last observation carried forward (LOCF).
Time Frame: Baseline and up to end of study (planned at Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of predicted FVC
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
Percent of predicted FVC
  Day 8 | -0.33 (7.93) | 0.04 (7.32)
  Day 29 | -0.76 (8.70) | -1.05 (9.12)
  Day 42 | 0.92 (8.98) | -1.09 (9.46)
  Day 56 | 0.36 (7.45) | -1.16 (9.83)
  Day 84 | -0.01 (7.57) | -1.99 (8.86)

4. Secondary Outcome: Time to Exacerbation With Antibiotic Intervention
Description: Acute exacerbation was defined according to the joint American Thoracic Society/European Respiratory Society criteria. For detailed information with regard to this definition of acute exacerbation, please refer to the detailed description in the protocol section. The time to an acute exacerbation with antibiotic intervention was determined.
Time Frame: Up to end of study (planned at Day 84)
Population: Modified intent-to-treat (ITT) analyses were performed on all participants who had been randomized and received study drug. This population was identical to the ITT population of all randomized participants. NA: due to fewer than 25% of participants having an exacerbation
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
Days | NA [NA to NA] — NA: due to fewer than 25% of participants having an exacerbation | NA [NA to NA] — NA: due to fewer than 25% of participants having an exacerbation

5. Secondary Outcome: Effect of Ciprofloxacin Inhale Treatment on Health-related Quality of Life (HRQoL) as Measured by the Saint George's Respiratory Questionnaire (SGRQ), Total Score
Description: Participants completed the Saint George's Respiratory Questionnaire (SGRQ). They were assured that all data would be treated confidentially and that the answers would not have any influence on study drug treatment. Participants completed the questionnaires on their own in a quiet area, without discussing them with study staff or accompanying persons (e.g. friends or relatives) and before being seen by the clinician. The score ranges from 0 to 100 with 100 being the worst possible score.
Time Frame: Up to end of study (planned at Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
Scores on a scale
  Day 1 | 43.8 (20.3) | 44.7 (18.1)
  Day 29 | 41.5 (21.0) | 44.8 (19.8)
  Day 56 | 40.6 (20.9) | 44.1 (18.6)
  Day 84 | 40.6 (18.1) | 41.6 (17.0)

6. Secondary Outcome: Effect of Ciprofloxacin Inhale Treatment on Health-related Quality of Life (HRQoL) as Measured by Chronic Respiratory Questionnaire - Self Administered Standardized (CRQ-SAS)
Description: Participants completed the Chronic Respiratory Questionnaire - Self Administered Standardized (CRQ-SAS). They were assured that all data would be treated confidentially and that the answers would not have any influence on study drug treatment. Participants completed the questionnaires on their own in a quiet area, without discussing them with study staff or accompanying persons (e.g. friends or relatives) and before being seen by the clinician. The score ranges between 1 and 7, 1 being the worst possible score.
Time Frame: Up to end of study (planned at Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Total score on a scale
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
Total score on a scale
  Day 1 | 4.88 (1.20) | 4.96 (0.98)
  Day 29 | 4.99 (1.21) | 4.93 (1.21)
  Day 56 | 4.94 (1.29) | 4.91 (1.16)
  Day 84 | 5.01 (1.21) | 4.99 (1.06)

7. Secondary Outcome: Change From Baseline in High Sensitive C-reactive Protein (hsCRP)
Description: High sensitive C-reactive protein (hsCRP) was determined from safety blood samples. Missing or invalid values were replaced with the last valid value available.
Time Frame: Baseline and up to Day 42
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
mg/L
  Day 8 | -0.43 [-4.10 to 0.40] | -0.19 [-2.48 to -0.19]
  Day 29 | 0 [-3.50 to 1.90] | 0 [-1.92 to 3.10]
  Day 42 | -0.16 [-4.40 to 1.91] | 0.12 [-2.07 to 3.10]

8. Secondary Outcome: Change From Baseline in Absolute Neutrophil Count (ANC)
Description: Absolute neutrophil count (ANC) was determined from safety blood samples. Missing or invalid values were replaced with the last valid value available.
Time Frame: Baseline and up to Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: giga/L
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
giga/L
  Day 8 | -0.35 (1.59) | -0.03 (1.45)
  Day 29 | -0.36 (1.69) | 0.59 (1.97)
  Day 42 | -0.28 (1.70) | 0.24 (2.21)

9. Secondary Outcome: 24-hour Sputum Volume
Description: Participants were asked to start 24-hour sputum collection samples 24 hours before coming for the respective study visit. The volume of the completed sample was determined.
Time Frame: Up to end of study (planned at Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
mL
  Day 1 | 24.9 (23.6) | 30.2 (25.2)
  Day 8 | 18.9 (22.2) | 30.0 (24.1)
  Day 29 | 20.5 (25.3) | 27.3 (32.5)
  Day 42 | 21.1 (24.7) | 22.8 (21.1)
  Day 56 | 19.6 (24.8) | 22.0 (24.8)
  Day 84 | 23.6 (28.9) | 25.9 (22.9)

10. Secondary Outcome: 24-hour Sputum Color (Percentage of Participants With Non-clear Sputum)
Description: Participants were asked to start 24-hour sputum collection samples 24 hours before coming for the respective study visit. Sputum color was assessed as either 'clear', or as 'yellow', 'green' or 'rust', or an assessment of 'no sputum' was made.
Time Frame: Up to end of study (planned at Day 84)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
Percentage of participants
  Day 1 | 91.7 | 88.9
  Day 8 | 73.2 | 94.9
  Day 29 | 75.5 | 82.7
  Day 42 | 72.8 | 88.4
  Day 56 | 75.0 | 86.5
  Day 84 | 66.6 | 72.8

11. Secondary Outcome: Microbiological Response of Cipro Inhale Per Participant
Description: Microbiological response was defined as reduction in bacterial load or eradication (measured as the percentage of participants with positive culture). Missing values were not imputed.
Time Frame: Up to end of study (planned at Day 84)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
Percentage of participants
  Day 1 | 100.0 | 100.0
  Day 8 | 52.4 | 88.2
  Day 29 | 65.0 | 91.8
  Day 42 | 83.3 | 86.8
  Day 56 | 87.1 | 96.4
  Day 84 | 85.2 | 92.0

12. Secondary Outcome: Microbiological Response of Cipro Inhale Per Pathogen
Description: Microbiological response was defined as reduction in bacterial load or eradication (measured as the number of participants with positive culture). Missing values were not imputed. Pathogens analyzed: Staphylococcus aureus, Streptococcus pneumoniae, Escherichia coli, Klebsiella pneumoniae, Klebsiella oxytoca, Proteus mirabilis, Serratia marcescens, Pseudomonas aeruginosa, mucoid, Pseudomonas aeruginosa, non mucoid, Stenotrophomonas maltophilia, Achromobacter xylosoxydans, Moraxella catarrhalis, Haemophilus influenzae
Time Frame: Up to end of study (planned at Day 84)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
Participants
  S. aureus Day 1 | 8 | 17
  S. aureus Day 8 | 4 | 7
  S. aureus Day 29 | 5 | 10
  S. aureus Day 42 | 6 | 9
  S. aureus Day 56 | 8 | 5
  S. aureus Day 84 | 5 | 5
  S. pneumoniae Day 1 | 7 | 2
  S. pneumoniae Day 8 | 2 | 4
  S. pneumoniae Day 29 | 0 | 4
  S. pneumoniae Day 42 | 3 | 1
  S. pneumoniae Day 56 | 1 | 2
  S. pneumoniae Day 84 | 1 | 1
  E. coli Day 1 | 2 | 2
  E. coli Day 8 | 2 | 2
  E. coli Day 29 | 2 | 1
  E. coli Day 42 | 0 | 1
  E. coli Day 56 | 1 | 0
  E. coli Day 84 | 1 | 0
  K. pneumoniae Day 1 | 5 | 0
  K. pneumoniae Day 8 | 0 | 0
  K. pneumoniae Day 29 | 0 | 0
  K. pneumoniae Day 42 | 0 | 1
  K. pneumoniae Day 56 | 1 | 0
  K. pneumoniae Day 84 | 3 | 0
  K. oxytoca Day 1 | 3 | 2
  K. oxytoca Day 8 | 0 | 1
  K. oxytoca Day 29 | 0 | 2
  K. oxytoca Day 42 | 0 | 1
  K. oxytoca Day 56 | 0 | 1
  K. oxytoca Day 84 | 1 | 1
  P. mirabilis Day 1 | 3 | 4
  P. mirabilis Day 8 | 0 | 3
  P. mirabilis Day 29 | 0 | 1
  P. mirabilis Day 42 | 2 | 3
  P. mirabilis Day 56 | 2 | 2
  P. mirabilis Day 84 | 2 | 2
  S. marcescens Day 1 | 2 | 3
  S. marcescens Day 8 | 0 | 2
  S. marcescens Day 29 | 0 | 3
  S. marcescens Day 42 | 0 | 3
  S. marcescens Day 56 | 0 | 2
  S. marcescens Day 84 | 2 | 0
  P. aeruginosa, mucoid Day 1 | 12 | 16
  P. aeruginosa, mucoid Day 8 | 7 | 15
  P. aeruginosa, mucoid Day 29 | 9 | 16
  P. aeruginosa, mucoid Day 42 | 9 | 12
  P. aeruginosa, mucoid Day 56 | 6 | 6
  P. aeruginosa, mucoid Day 84 | 4 | 5
  P. aeruginosa, non mucoid Day 1 | 20 | 19
  P. aeruginosa, non mucoid Day 8 | 6 | 17
  P. aeruginosa, non mucoid Day 29 | 10 | 14
  P. aeruginosa, non mucoid Day 42 | 12 | 12
  P. aeruginosa, non mucoid Day 56 | 10 | 9
  P. aeruginosa, non mucoid Day 84 | 13 | 6
  S. maltophilia Day 1 | 2 | 3
  S. maltophilia Day 8 | 0 | 3
  S. maltophilia Day 29 | 2 | 3
  S. maltophilia Day 42 | 2 | 1
  S. maltophilia Day 56 | 4 | 3
  S. maltophilia Day 84 | 1 | 1
  A. xylosoxydans Day 1 | 2 | 3
  A. xylosoxydans Day 8 | 2 | 2
  A. xylosoxydans Day 29 | 2 | 1
  A. xylosoxydans Day 42 | 2 | 0
  A. xylosoxydans Day 56 | 1 | 1
  A. xylosoxydans Day 84 | 0 | 2
  M. catarrhalis Day 1 | 5 | 3
  M. catarrhalis Day 8 | 0 | 3
  M. catarrhalis Day 29 | 0 | 6
  M. catarrhalis Day 42 | 1 | 2
  M. catarrhalis Day 56 | 1 | 2
  M. catarrhalis Day 84 | 1 | 2
  H. influenzae Day 1 | 14 | 16
  H. influenzae Day 8 | 1 | 12
  H. influenzae Day 29 | 1 | 11
  H. influenzae Day 42 | 1 | 7
  H. influenzae Day 56 | 3 | 8
  H. influenzae Day 84 | 4 | 8

13. Secondary Outcome: Emergence of New Potential Respiratory Pathogens
Description: The emergence of new potential respiratory pathogens was evaluated using microbiological analysis. Evaluated was the cumulative number of participants with first appearance of new potential respiratory antigens at each time point. In some cases, participants attended the end of study visit later than Day 84 (up to Day 88).
Time Frame: Up to end of study (planned at Day 84)
Population: as for outcome 1
Measure: Number; unit: Cumulative participants
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
Cumulative participants
  Day 4 | 1 | 0
  Day 5 | 1 | 2
  Day 7 | 2 | 2
  Day 8 | 7 | 8
  Day 9 | 7 | 10
  Day 10 | 7 | 11
  Day 14 | 7 | 12
  Day 15 | 7 | 13
  Day 28 | 7 | 14
  Day 29 | 12 | 24
  Day 30 | 14 | 30
  Day 36 | 15 | 30
  Day 39 | 16 | 31
  Day 42 | 18 | 33
  Day 43 | 21 | 38
  Day 44 | 25 | 40
  Day 45 | 26 | 41
  Day 57 | 29 | 45
  Day 58 | 29 | 46
  Day 59 | 30 | 47
  Day 78 | 31 | 47
  Day 83 | 32 | 47
  Day 84 | 33 | 47
  Day 85 | 38 | 53
  Day 86 | 41 | 54
  Day 88 | 43 | 54

14. Secondary Outcome: Emergence of Resistance Among Baseline Pathogens
Description: The emergence of resistance (at least two-fold increase of Minimal inhibitory concentration, MIC, vs. baseline values) probably or possibly related to study medication among baseline pathogens was evaluated using microbiological analysis.
Time Frame: Up to end of study (planned at Day 84)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
Participants
  Emergence (>= 2* increase of MIC) | 7 | 1
  Sustained (>= 2* increase of MIC until end) | 1 | 0
  Transient (Increase in MIC with normalization) | 5 | 1
  Insufficient follow up | 1 | 0

15. Other Pre Specified Outcome: Change From Baseline in Total Bacterial Load in the Sputum
Description: Total bacterial load was determined in sputum collected before the inhalation of study drug. Sputum samples were either provided by the participant during the respective study visit, or participants had to bring a sputum sample that had been produced within the 4 hours prior to the visit. Induced sputum samples could be collected if the participant was unable to produce a spontaneously expectorated sputum sample of > 2 mL on Day 8. Imputation method: last observation carried forward (LOCF). CFU: colony forming units, log10: decadic logarithm
Time Frame: Baseline and up to end of study (planned at Day 84)
Population: Modified intent-to-treat (ITT) analyses were performed on all participants who had been randomized and received study drug. This population was identical to the ITT population of all randomized participants. Decadic logarithm of colony forming units (CFUs) per gram sputum
Measure: Mean (Standard Deviation); unit: log10 of CFU per gram sputum
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Number analyzed (Participants) | 60 | 64
log10 of CFU per gram sputum
  Day 8 | -2.87 (3.39) | -0.20 (2.15)
  Day 42 | -1.86 (3.06) | -0.31 (2.08)
  Day 56 | -1.86 (3.11) | -0.21 (1.89)
  Day 84 | -1.37 (3.17) | -0.24 (1.77)

ADVERSE EVENTS:
Arm/Group | Ciprofloxacin Inhale (BAYQ3939) | Placebo
Serious Adverse Events (participants affected / at risk) | 4/60 | 6/64
Other Adverse Events (participants affected / at risk) | 38/60 | 36/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciprofloxacin Inhale (BAYQ3939) (N=60) | Placebo (N=64)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bronchiectasis (Infections and infestations) | 1 (1) | 5 (6)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciprofloxacin Inhale (BAYQ3939) (N=60) | Placebo (N=64)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Product taste abnormal (General disorders) | 8 (8) | 7 (7)
Bronchiectasis (Infections and infestations) | 22 (24) | 22 (23)
Dysgeusia (Nervous system disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 6 (7) | 6 (8)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must send a draft manuscript of the publication or abstract to the sponsor 30 days in advance of submission in order to obtain written approval prior to submission of the final version for publication. This will be reviewed promptly and approval will not be withheld unreasonably. In case of a difference of opinion, the contents of the publication will be discussed in order to find a solution that satisfies both parties.